CLINICAL TRIAL: NCT05110092
Title: Breathing-based Leg Resistance Exercise Improves Wound Healing, Blood Sugar and Quality of Life for Diabetic Foot Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016-08-006B
Record Dates: First submitted 2021-09-06; First posted 2021-11-05 (Actual); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Diabetic Foot; Resistance Exercise; Wound Healing; Hyperglycemia; Quality of Life
MeSH Terms: conditions — Diabetic Foot; Hyperglycemia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The exercise group (Experimental): The exercise group received usual care and breathing-based leg resistance exercise program for 12 weeks.
  Interventions: Behavioral: leg resistance combined with breathing exercise training
- The control groups (No Intervention): The control group received usual care

INTERVENTIONS:
Behavioral: leg resistance combined with breathing exercise training — The exercise group was provided breathing and leg resistance exercise manuals. The exercise involved 5 minutes of abdominal breathing in a relaxed sitting position, followed by 10 minutes of leg resistance training.
  Arms: The exercise group

SUMMARY:
The purpose of the study was designed leg resistance training combined with breathing approach, and evaluated its effect on wound healing, blood sugar control and quality of life in type 2 diabetic patients with foot ulcers.

DETAILED DESCRIPTION:
A randomized controlled trial was used. type 2 diabetic patients who suffered from foot ulcers were recruited from one medical center of Northern Taiwan, and randomly assigned into the exercise or control group. The control group received usual care for diabetic foot. The exercise group received usual care and breathing-based leg resistance exercise program for 12 weeks. Outcomes were measured by wound healing area, the fasting of blood glucose, hemoglobin A1c (HbA1c), and the World Health Organization quality of life-BREF (WHOQOL-BREF) before the intervention as baseline, and the 4th, 8th and 12th weeks during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

* patients 20 years or older
* who were diagnosed with type 2 diabetic foot
* ulcers of Meggitt-Wagner Grade 1-2
* who were conscious and could perform the prescribed exercise.

Exclusion Criteria:

* peripheral arterial occlusion disease
* osteomyelitis
* inability to perform exercise as assessed by physicians.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2016-12-14 (Actual); Primary Completion 2021-11-11 (Estimated); Study Completion 2021-11-11 (Estimated)

PRIMARY OUTCOMES:
wound healing | during 12 weeks the intervention period.
  wound size(cm2)
blood sugar control-fasting blood sugar | during 12 weeks the intervention period.
  fasting blood sugar(mg/dl ) using a blood glucose meter
quality of life measured by the World Health Organization Quality of Life-BREF | during 12 weeks the intervention period.
  Quality of life was measured using the World Health Organization Quality of Life-BREF (WHOQOL-BREF) in the Taiwan version
blood sugar control-HbA1c | during 12 weeks the intervention period.
  The levels of hemoglobin A1c (%)(HbA1c) were monitored blood sugar in the long term